CLINICAL TRIAL: NCT04190771
Title: Efficacy of a Multicomponent Intervention for Fibromyalgia Based on Physical Activity, Psychological Support, and Nature Exposure (NAT-FM)
Brief Title: Efficacy of NAT-FM Treatment for Fibromyalgia
Acronym: NAT-FM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Parc Sanitari Sant Joan de Déu (Other); Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAT-FM
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Fibromyalgia
Keywords: multicomponent treatment; Nature therapy; Mindfulness; Physical therapy; Pain Neuroscience Education (PNE)
MeSH Terms: conditions — Fibromyalgia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Single-blind, parallel-group, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + multicomponent treatment NAT-FM (Experimental): NAT-FM is a multicomponent non-pharmacological program based on mindfulness ingredients, pain neuroscience education, and nature exposure. NAT-FM is conceived as an add-on therapy.
  Interventions: Behavioral: TAU + multicomponent treatment NAT-FM; Behavioral: Treatment as Usual (TAU)
- Treatment as Usual (TAU) (Active Comparator): Standard Care. Although there is no treatment considered as the gold standard for fibromyalgia, the standard treatment is usually mainly pharmacological and conforms to the symptomatic profile of each patient.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: TAU + multicomponent treatment NAT-FM — Group treatment protocol of 12 weekly 120 minute sessions. All sessions include the following ingredients (approx. in the same order):
  * Pain neuroscience education (30 min.)
  * Cognitive restructuring (30 min.)
  * Mindfulness techniques (30 min.)
  * Physical exercise in a natural environment / nature exposure (30 min.) Treatment as Usual (TAU) Standard pharmacological treatment usually provided to patients with fibromyalgia.
  Arms: TAU + multicomponent treatment NAT-FM
Behavioral: Treatment as Usual (TAU) — Standard pharmacological treatment usually provided to patients with fibromyalgia.

SUMMARY:
The main objective of this study is to analyse the efficacy of the NAT-FM multicomponent treatment program as coadjuvant of treatment-as-usual (TAU) compared to TAU alone.

In this Randomized Controlled Trial (RCT), in addition to evaluating the clinical effects of NAT-FM treatment in the short- and long-term, the research team will seek to identify relevant moderators and mediators of clinical change.

DETAILED DESCRIPTION:
* This is a two-arm RCT focused on the safety and potential efficacy of the multicomponent program NAT-FM as coadjuvant of treatment-as-usual (TAU) vs. TAU alone.
* NAT-FM combines Classical Structural Assessment (CSA) and Ecological Momentary Assessment (EMA) to obtain more reliable information about the dynamics of the variables to be evaluated, to record the affective and cognitive impact of each activity, and to explore its potential delivery in real-world clinical practice.
* The main hypothesis is that improvement on functional impairment of patients with fibromyalgia can be achieved by the direct intervention on mechanisms such as self-efficacy and pain catastrophizing.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 to 75 years-old.
* 1990 American College of Rheumatology (ACR) classification criteria + the 2011 modified ACR diagnostic criteria for fibromyalgia
* Able to understand Spanish and accept to participate in the study.

Exclusion Criteria:

* Participating in concurrent or past RCTs (previous year).
* Comorbidity with severe mental disorders (i.e. psychosis) or neurodegenerative diseases (i.e. Alzheimer) that that would limit the ability of the patient to participate in the RCT.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQR) | Through study completion, an average of 9 months
  The FIQR comprises three dimensions: physical dysfunction (scores from 0 to 30), overall impact (scores from 0 to 20), and intensity of the symptoms (scores from 0 to 50) is used to measure the impact generated by FM during the last week. It consists of 21 items, which are answered on a numerical rating scale of 11 points (from 0 to 10). Total scores can range from 0 to 100, with higher scores reflecting greater deterioration.

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK-11) | Through study completion, an average of 9 months
  TSK-11 is used to assess fear of pain and movement. It consists of 11 items, which are answered on a Likert scale of 4 points. Total scores of each scale range from 11 to 44, where higher scores indicate a greater fear of pain and movement.
Hospital Anxiety and Depression Scale (HADS) | Through study completion, an average of 9 months
  HADS is used to quantify the severity of anxiety and depression symptoms. It consists of two dimensions (anxiety and depression) of 7 items each responding on a Likert scale of 4 points. Total scores of each scale (HADS-A and HADS-D) range from 0 to 21, where higher scores indicate greater severity of symptoms.
Pain Catastrophizing Scale (PCS) | Through study completion, an average of 9 months
  PCS is used to evaluate catastrophic thoughts associated with pain. It consists of three dimensions (rumination, magnification, and helplessness) of 13 items in total, which are answered on a Likert scale of 5 points. Total scores on each scale range from 0 to 52, with higher scores indicating more catastrophic thoughts.
Perceived Stress Scale (PSS) | Through study completion, an average of 9 months
  PSS is used to evaluate the stress perceived by people during the last month. This study will use a 4 item version. The response format of this scale is 5-point Likert type. Total scores range from 0 to 16, with higher scores indicating greater perceived stress.
Personal Perceived Competence Scale (PPCS) | Through study completion, an average of 9 months
  PPCS is used to measure perceived competence. It consists of 8 items that are answered on a 6-point Likert scale. Total scores of each scale range from 8 to 48, with higher scores indicating greater perceived competence.
Rosenberg Self-Esteem Scale (RSES) | Through study completion, an average of 9 months
  RSES is used to measure self-esteem. It consists of 10 items that are answered on a Likert scale of 4 points. Total scores of each scale range from 10 to 40, where higher scores indicate higher self-esteem.
Cognitive Emotion Regulation Questionnaire (CERQ) | Through study completion, an average of 9 months
  CERQ is used to assess individual differences in the cognitive regulation of emotions. The instrument measures nine 2-item dimensions (self-blame, blaming others, acceptance, refocusing on planning, positive refocusing, rumination, positive reappraisal, putting into perspective, and catastrophizing). This study will use the short version of 18 items. Responses are given on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). Total scores for each dimension range from 2 to 10, with the highest scores indicating the specific cognitive strategy most used.
Positive and Negative Affect Schedule (PANAS) | Through study completion, an average of 9 months
  PANAS is used to evaluate positive and negative affect. It consists of two dimensions (positive affect and negative affect) of 10 items each answered on a Likert scale of 5 points. Total scores of each scale range from 10 to 50, where higher scores indicate a greater presence of the specific affectivity.
Ecological Momentary Assessment (EMA) | Through intervention completion, an average of 3 months
  Use of a commercial app used to assess daily (four times a day) the level of pain, fatigue, pain catastrophism during the monitoring period.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Marsal Barril, PhD, Study Chair — Vall d'Hebrón Hospital
Locations (1):
- Vall d'Hebrón Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No